CLINICAL TRIAL: NCT07402863
Title: Self-Guided Resilience-Building Energy Management to Enhance Well-being Intervention for People With Systemic Sclerosis: A Feasibility Study
Brief Title: Self-Guided Resilience-Building Energy Management to Enhance Well-being (RENEW) Intervention for People With Systemic Sclerosis (SSc)
Acronym: RENEW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Shepherd Center, Atlanta GA (Other); National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Susan Murphy, Title Professor of Physical Medicine and Rehabilitation, Research Professor, Institute of Gerontology and Professor of Internal Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUM00266174; SHEP-20-0010 (Other Grant/Funding Number: Shepherd Center, Inc., Atlanta, Georgia); 90DPHF0004 (Other Grant/Funding Number: National Institute on Disability, Independent Living and Rehabilitation Research)
Record Dates: First submitted 2026-01-21; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RENEW (Experimental): Individuals with SSc who are interested and eligible will undergo an informed consent process and will be given access to the RENEW program via the app
  Interventions: Device: RENEW

INTERVENTIONS:
Device: RENEW — The RENEW program is 12-week program where participants are asked to access the app and set and track weekly healthy goals.

SUMMARY:
The goal of this clinical trial is to gather information on the RENEW app used by people with scleroderma. Specifically, the researchers want to learn more about RENEW by collecting information about the rates of recruitment, retention of study participants information about study completion, and time spent accessing the app content.

DETAILED DESCRIPTION:
RENEW is Institutional Review Board approved as a non-significant risk device but it not subject to 510(k) and therefore not regulated by the FDA.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of systemic sclerosis including: diffuse cutaneous SSc, limited cutaneous SSc, overlap, or SINE
* Have access to a reliable, internet-connected device (e.g. smartphone or tablet)
* Be able to read, speak, and understand English
* Participants need to report a score of at least 4 on a scale of 0 - 10 of fatigue severity, a cut-off for at least moderate fatigue in other fatiguing conditions1

Exclusion Criteria:

* Complex, unstable health issues that would preclude full participation in the study
* Planning to start new treatment for fatigue, pain, mood during the study period
* Previous experience with RENEW app or past participant of RENEW

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2025-01-28 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
Feasibility based on study recruitment rate | 12 weeks
  Number of participants enrolled (over 3 months) divided by the number of individuals who were eligible to participate
Feasibility based on study retention | 12 weeks
  Number of participants who complete the study

SECONDARY OUTCOMES:
RENEW participation - website | 12 weeks
  Reported as the number of minutes spent accessing the RENEW app
Acceptability | 12 weeks
  Assessed using the 12-week feedback questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Susan Murphy, ScD, OTR, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No